CLINICAL TRIAL: NCT00106860
Title: A Long-Term, Open Label, Safety and Efficacy Study of an Experimental Medication in Adults With Generalized Anxiety Disorder (GAD)
Brief Title: A Long-Term Study Continuing on From Study 04-001-01 of an Experimental Medication in Adults With Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-003
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2008-01

CONDITIONS: Anxiety Disorder
Keywords: Anxiety; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

INTERVENTIONS:
Drug: a benzodiazepine drug

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of the experimental drug, a benzodiazepine drug, in long-term use and the effects on quality of life, social and occupational functioning, sleep, and daytime sedation in subjects with anxiety disorder.

DETAILED DESCRIPTION:
This trial is a long-term, open label, safety and efficacy study of an experimental medication in adults with Generalized Anxiety Disorder (GAD). To enroll in this study, investigators and patients must have first participated in Jazz Pharmaceuticals, Inc. Protocol 04-001-01. The study is designed for four stages that should last a total of 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Complete Study 04-001-01
* Able to take the medication for 9 months
* Understand and sign the Informed Consent
* Comply with all study-related procedures
* Women of child bearing potential must have a confirmed negative urine pregnancy test
* Lack of clinically significant abnormalities in health

Exclusion Criteria:

* Experienced any SAEs (serious adverse events) that were related or possibly related to study drug during participation in Study 04-001-01
* Early termination from study 04-001-01
* Any new condition that could interfere with the evaluation of the subject, interpretation of safety data, or compliance with the protocol requirements
* Experiencing AEs (adverse events) such that in the opinion of the investigator, per protocol, study drug administration or safe participation in this study would be precluded.
* Taken any disallowed medications noted in Study 04-001-01 between the completion of Study 04-001-01 and entry into this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158
Dates: Start 2005-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Assessment (over 37 additional weeks following the double-blind study) of the safety of the experimental drug in long-term use in subjects with Generalized Anxiety Disorder (GAD)

SECONDARY OUTCOMES:
Evaluate the long-term efficacy of open-label study of the experimental drug in subjects with GAD
Assessment of the long-term effects on the quality of life, social and occupational functioning, sleep, and daytime sedation in subjects with GAD

CONTACTS AND LOCATIONS:
Overall Officials: Murray Stein, MD, Study Chair — University of California, San Diego
Locations (13):
- United States (13):
  - Florida Clinical Research Center, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Meridien Research, St. Petersburg, Florida
  - CNS Research Institute (CRI), Clementon, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology and NeuroscienceCenter of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Research, Inc., Eugene, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - CNS Research Institute (CRI), Philadelphia, Pennsylvania
  - Future Search Trials, Austin, Texas
  - Comprehensive Neuroscience of Northern Virginia, Falls Church, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington